CLINICAL TRIAL: NCT03893214
Title: Virtual Reality Exposure Therapy for Acrophobia in a Single Session Design and the Role of Respiration for Fear Extinction
Brief Title: Single Session Virtual Reality Therapy in Acrophobia - and the Role of Respiration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Witten/Herdecke (Other)
Collaborators: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Prof. Dr. Johannes Michalak, Full Professor, University of Witten/Herdecke
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VRAcro
Record Dates: First submitted 2019-03-14; First posted 2019-03-28 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Acrophobia
Keywords: virtual reality exposure therapy; waitlist control design; single session exposure; emotion-driven behavior; respiration
MeSH Terms: conditions — Acrophobia; Respiratory Aspiration | interventions — Motion Pictures

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two conditions (virtual reality vs. waitlist control) for the initial phase. In the second phase the waitlist control group receives the virtual reality exposure while the other group does not receive a second intervention.
Masking Description: All roles are aware of the fact that the virtual reality exposure is the primary intervention. No information is given to the participant about the impact of the "video" in the waitlist control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Virtual reality exposure for acrophobia - this arm receives the virtual reality exposure intervention in the initial phase and has a four-week follow-up assessment.
  Interventions: Behavioral: virtual reality exposure for acrophobia
- waitlist control group (Placebo Comparator): This arm watches a movie in the initial phase in order to control for effects of behavioral approach test that is done before and after the intervention and for time effects. In the second phase after four weeks, this arm receives the virtual reality exposure after collection of outcome measures.
  Interventions: Behavioral: virtual reality exposure for acrophobia; Behavioral: movie

INTERVENTIONS:
Behavioral: virtual reality exposure for acrophobia — The setting of the virtual reality is the "Gasometer Oberhausen", Europe's largest disc-type gas container which is one of the most famous high buildings in the area. After a baseline phase, participants will undergo a gradual exposure. Participants will first look up to the building and then be guided upstairs to have an exposure phase on 11 floors. On the highest floor they will walk around a gallery. In the end, there will be a recovery phase.
Behavioral: movie — Participants will watch a movie without height content for the same amount of time as the virtual reality exposure will need.
  Arms: waitlist control group

SUMMARY:
In recent years, in the treatment of phobias, exposure therapy in virtual reality is becoming more and more popular as an alternative for in-vivo exposure. Effectiveness of virtual reality exposure therapy (VRET) is comparable to in-vivo exposure therapy, though several characteristics of the VRET have an impact on the outcome of the therapy (e.g., immersion into the virtual environment (VE), familiarity with the VE). Additionally, the use of VRET varies from multiple exposure sessions to single-session VRET. Single-session therapy has an economic advantage and in in-vivo, post therapy outcomes show good results. In virtual reality, the assessment of outcome post therapy and in follow-up of single-session therapies is still needed for an evaluation of this approach. As an outcome measure, behavioral assessments are especially relevant for effectiveness studies as in fear of heights it is closer to the individual's life to know how high they voluntarily go up a building than to have hypothetical self-report questionnaire results.

Much research has been conducted on physiological correlates of the subjective experience of fear in exposure therapy as they are assumed to be a prerequisite for effective exposure treatment. Skin conductance level (SCL) and heart rate can be used for objective manipulation checks of exposure therapy. SCL is found to increase during fearful situations independent of setting while heart rate only increases during in-vivo exposure. Contrary to heart rate, heart rate variability (HRV) is not thoroughly studied in VRET yet. HRV is associated with the adaptability of an organism to new environments and cognitive functioning. High Frequency HRV is found to be reduced in individuals with mental disorders, and positive and negative mood inductions lead to differential HRV responses overall.

Respiration is a well-studied correlate of emotional experience and especially of the experience of fear and anxiety. In a series of experiments, it was found that sighing is tightly associated with relief in or after fearful or stressful situations and might become maladaptive when used disproportionally often. This study shows that respiration parameters have an impact on the handling of fearful situations in a reciprocal way. On the one hand, fear leads to an increased respiration rate and sigh rate while on the other hand, an altered sigh rate or respiration rate might have an impact on the experience of fear and be used as a defensive reaction to a fearful situation. As such, specific respiration patterns might act as emotion-driven behaviors (EDB). EDBs are responses to emotions that result in a short-term reduction of a negative state while in long-term support the maintenance of the phobia.

The aim of this study is to examine the effectiveness of a single-session VRET for acrophobia with a multimethod outcome design. Familiarity of the setting will be high with the use of a well-known tower in this area. Immersion into the VE will be assessed with a presence questionnaire. For a manipulation check, physiological data will be assessed, i.e., SCL, heart rate and HRV. Primary outcome measure will be a behavioral approach test (BAT) as behavioral assessment. Additionally, after four weeks, a follow-up assessment will investigate the stability of the effectiveness of the VRET in comparison to a waitlist control group. A second aim of this study is to investigate the impact of respiration as an EDB on the effectiveness of an exposure therapy. Therefore, the association between respiration and outcome of the VRET will be analyzed.

Hypothesis 1: Participants in the VRET condition show less height avoidance in the BAT after the intervention than participants in the control condition.

Hypothesis 2: Participants in the VRET condition show less height avoidance in the BAT in a four-week follow-up assessment than participants in the control condition.

Hypothesis 3: Participants in the VRET condition score significantly lower on the Acrophobia Questionnaire at follow-up than participants in the control condition.

Hypothesis 4: During the VRET, breath holding is used as EDB. Participants that hold their breath, profit less from the VRET than participants that do not hold their breath.

Hypothesis 5: During the VRET, sighing is used as EDB. Participants that sigh, profit less from the VRET than participants that do not sigh.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed acrophobia
* read, speak and write in German language

Exclusion Criteria:

* current panic disorder
* lifetime psychotic disorder
* current suicidality
* neurological disorder
* current substance use disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Equal gender distribution will be ensured because physiological processes and their impact on psychological processes can differ between men and women.
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Behavioral Approach Test Post | Within 1 hour after treatment /placebo intervention
  Participants are asked to walk up fire exit stairs of the university building where the treatment is applied. The number of steps upstairs is counted as dependent measure.
Behavioral Approach Test Follow-up | Four weeks +/- 3 day after the treatment / placebo intervention
  Participants are asked to walk up fire exit stairs of the university building where the treatment is applied. The number of steps upstairs is counted as dependent measure.

SECONDARY OUTCOMES:
Acrophobia Questionnaire Follow-up | Four weeks +/- 3 day after the treatment / placebo intervention
  Questionnaire by Cohen (1977); The scale ranges from 0 - not at all frightening to 6 - very frightening with a higher score indicating more anxiety. A total maximum score is 120 and minimum score 0.
Sigh Rate | During virtual reality exposure session, at baseline (1; 5 minutes), on each floor of the tower (2-14; 3 minutes, in total 39 minutes) and in recovery phase (15; 5 minutes)
  Measured with inductive plethysmography and analyzed via ANSLAB
Number of Apnoeas | During virtual reality exposure session, at baseline (1; 5 minutes), on each floor of the tower (2-14; 3 minutes, in total 39 minutes) and in recovery phase (15; 5 minutes)
  Pauses after inspiration and expiration longer than 5 seconds, measured with inductive plethysmography and analyzed via ANSLAB
Respiration Rate | During virtual reality exposure session, at baseline (1; 5 minutes), on each floor of the tower (2-14; 3 minutes, in total 39 minutes) and in recovery phase (15; 5 minutes)
  Measured with inductive plethysmography and analyzed via ANSLAB
Respiratory Instability | During virtual reality exposure session, at baseline (1; 5 minutes), on each floor of the tower (2-14; 3 minutes, in total 39 minutes) and in recovery phase (15; 5 minutes)
  Measured with inductive plethysmography and analyzed via ANSLAB
Subjective Units of Discomfort Change | During virtual reality exposure session, at baseline (1; minute 1), on each floor of the tower (2-14; between minute 6 and 44) and in recovery phase (15; minute 50)
  Participants are asked how fearful they are on a scale from 0 to 10. Original scale by Wolpe & Lazarus (1966)
Heart Rate | During virtual reality exposure session, at baseline (1; 5 minutes), on each floor of the tower (2-14; 3 minutes, in total 39 minutes) and in recovery phase (15; 5 minutes)
  Measured with Electrocardiogram and analyzed via ANSLAB
Heart Rate Variability | During virtual reality exposure session, at baseline (1; 5 minutes), on each floor of the tower (2-14; 3 minutes, in total 39 minutes) and in recovery phase (15; 5 minutes)
  Measured with Electrocardiogram and analyzed via ANSLAB
Skin conductance level | During virtual reality exposure session, at baseline (1; 5 minutes), on each floor of the tower (2-14; 3 minutes, in total 39 minutes) and in recovery phase (15; 5 minutes)
  Skin conductance is recorded continuously with two electrodes placed on the medial phalanxes of the index and middle fingers of the nondominant hand.
Video recording | During virtual reality exposure session, at baseline (1; 5 minutes), on each floor of the tower (2-14; 3 minutes, in total 39 minutes) and in recovery phase (15; 5 minutes)
  A rating system for signs of muscular tension during virtual reality exposure will be designed. Therefore, in a first step it will be assessed whether signs of muscular tension are visible overall. In a second step, all signs from up to 10 randomly picked participants will be noted from two different raters in order to design a rating scale. This scale will then be applied to the rest of the participants by 2 independent raters and finally correlated with the post outcome measures and follow-up outcome measures.

OTHER OUTCOMES:
Anxiety Sensitivity Scale 3 Pre | Right before the randomization to treatment / placebo condition - within 1 hour before intervention / placebo intervention
  Questionnaire by Kemper, Ziegler & Taylor (2009); Scale ranges from 0 - very little to 4 - very much; a total maximum score is 64 and a minimum 0 with a higher score indicating more anxiety sensitivity.
Anxiety Sensitivity Scale 3 Follow-up | Four weeks +/- 3 day after the treatment / placebo intervention
  Questionnaire by Kemper, Ziegler & Taylor (2009); Scale ranges from 0 - very little to 4 - very much; a total maximum score is 64 and a minimum 0 with a higher score indicating more anxiety sensitivity.
Self-Evaluation of Breathing Questionnaire Follow-up | Four weeks +/- 3 day after the treatment / placebo intervention
  Questionnaire by Courtney & Greenwood (2009) - translated with backtranslation by the author. The scale ranges from 0 - never to 3 - very often with a higher score indicating more breathing dirsturbances. A total maximum score is 75 and minimum 0.
Self-Evaluation of Breathing Questionnaire Pre | Right before the randomization to treatment / placebo condition - within 1 hour before intervention / placebo intervention
  Questionnaire by Courtney & Greenwood (2009) - translated with backtranslation by the author. The scale ranges from 0 - never to 3 - very often with a higher score indicating more breathing dirsturbances. A total maximum score is 75 and minimum 0.
Beck Depression Inventory II Follow-up | Four weeks +/- 3 day after the treatment / placebo intervention
  Questionnaire by Beck, Steer & Brown (2001), German version by Hautzinger, Keller & Kühner (2009). The scale ranges from 0 to 3 with a higher score indicating more depressive symptoms. A total maximum score is 60 and minimum score 0.
Beck Depression Inventory II Pre | Right before the randomization to treatment / placebo condition - within 1 hour before intervention / placebo intervention
  Questionnaire by Beck, Steer & Brown (2001), German version by Hautzinger, Keller & Kühner (2009). The scale ranges from 0 to 3 with a higher score indicating more depressive symptoms. A total maximum score is 60 and minimum score 0.
Igroup Presence Questionnaire | Within 30 minutes after virtual reality exposure (treatment)
  Questionnaire by Schubert, Friedmann & Regenbrecht (2001) to measure the feeling of presence in the virtual reality. Scale ranges from -3 - not at all to +3 - a lot with a total maximum score of 42 and minimum -42. A higher scores indicates a higher feeling of presence in the virtual reality.
Simulator Sickness Questionnaire | Within 30 minutes after virtual reality exposure (treatment)
  Questionnaire by Kennedy, Lane, Berbaum & Lilienthal (1993) to measure simulator sickness in the virtual reality. Scale ranges from 0 - not at all to 3 - strongly with a total maximum score of 48 and minimum 0. A higher scores indicates a higher feeling of simulator sickness in the virtual reality.
Mini-DIPS (Diagnostisches Interview bei psychischen Störungen; english: diagnostic interview of mental disorders) | Within a month before the treatment / placebo intervention
  Diagnostic interview to diagnose acrophobia and to exclude panic disorder. Interview by Margraf & Cwik (2017)
Behavioral Approach Test Pre | Right before the randomization to treatment / placebo condition - within 1 hour before treatment or placebo intervention
  Participants are asked to walk up fire exit stairs of the university building where the treatment is applied. The number of steps upstairs is counted as dependent measure. BAT pre is assessed in order to ensure an effective randomization.
Acrophobia Questionnaire Pre | Within a month before the treatment / placebo intervention
  Questionnaire by Cohen (1977); Screening for people with fear of hights and in order to ensure an effective randomization. The scale ranges from 0 - not at all frightening to 6 - very frightening with a higher score indicating more anxiety. A total maximum score is 120 and minimum score 0.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Adolph, PhD, Principal Investigator — Ruhr-University Bochum

IPD SHARING:
Plan to Share IPD: Yes
All collected de-identified individual participant data will be shared with other researchers.
Supporting Information: Study Protocol, ICF
Time Frame: All data will become available for six months with publication.
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Background] Barlow DH, Farchione TJ, Bullis JR, Gallagher MW, Murray-Latin H, Sauer-Zavala S, Bentley KH, Thompson-Hollands J, Conklin LR, Boswell JF, Ametaj A, Carl JR, Boettcher HT, Cassiello-Robbins C. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders Compared With Diagnosis-Specific Protocols for Anxiety Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Sep 1;74(9):875-884. doi: 10.1001/jamapsychiatry.2017.2164. PMID 28768327
- [Background] Beauchaine TP, Thayer JF. Heart rate variability as a transdiagnostic biomarker of psychopathology. Int J Psychophysiol. 2015 Nov;98(2 Pt 2):338-350. doi: 10.1016/j.ijpsycho.2015.08.004. Epub 2015 Aug 11. PMID 26272488
- [Background] Benke C, Hamm AO, Pane-Farre CA. When dyspnea gets worse: Suffocation fear and the dynamics of defensive respiratory responses to increasing interoceptive threat. Psychophysiology. 2017 Sep;54(9):1266-1283. doi: 10.1111/psyp.12881. Epub 2017 May 3. PMID 28466488
- [Background] Carl E, Stein AT, Levihn-Coon A, Pogue JR, Rothbaum B, Emmelkamp P, Asmundson GJG, Carlbring P, Powers MB. Virtual reality exposure therapy for anxiety and related disorders: A meta-analysis of randomized controlled trials. J Anxiety Disord. 2019 Jan;61:27-36. doi: 10.1016/j.janxdis.2018.08.003. Epub 2018 Aug 10. PMID 30287083
- [Background] Cohen DC. Comparison of self-report and overt-behavioral procedures for assessing acrophobia. Behavior Therapy 8(1): 17-23, 1977.
- [Background] Courtney R, Greenwood KM. Preliminary investigation of a measure of dysfunctional breathing symptoms: The Self Evaluation of Breathing Questionnaire (SEBQ). International Journal of Osteopathic Medicine 12(4): 121-127, 2009.
- [Background] Diemer J, Muhlberger A, Pauli P, Zwanzger P. Virtual reality exposure in anxiety disorders: impact on psychophysiological reactivity. World J Biol Psychiatry. 2014 Aug;15(6):427-42. doi: 10.3109/15622975.2014.892632. Epub 2014 Mar 25. PMID 24666248
- [Background] Hautzinger M, Keller F, Kühner C. BDI-II - Beck Depressions-Inventar Revision. London: Pearson, 2009.
- [Background] Jerath R, Crawford MW. How Does the Body Affect the Mind? Role of Cardiorespiratory Coherence in the Spectrum of Emotions. Adv Mind Body Med. 2015 Fall;29(4):4-16. PMID 26535473
- [Background] Kemper CJ, Ziegler M, Taylor S. Überprüfung der psychometrischen Qualität der deutschen Version des Angstsensitivitätsindex-3. Diagnostica 55(4): 223-233, 2009.
- [Background] Kennedy RS, Lane NE, Berbaum KS, Lilienthal MG. Simulator Sickness Questionnaire: An Enhanced Method for Quantifying Simulator Sickness. The International Journal of Aviation Psychology 3(3): 203-220, 1993.
- [Background] Kop WJ, Synowski SJ, Newell ME, Schmidt LA, Waldstein SR, Fox NA. Autonomic nervous system reactivity to positive and negative mood induction: the role of acute psychological responses and frontal electrocortical activity. Biol Psychol. 2011 Mar;86(3):230-8. doi: 10.1016/j.biopsycho.2010.12.003. Epub 2010 Dec 21. PMID 21182891
- [Background] Margraf J, Cwik JC. Mini-DIPS - Open Access - Diagnostisches Kurzinterview bei psychischen Störungen. 2017.
- [Background] Morina N, Ijntema H, Meyerbroker K, Emmelkamp PM. Can virtual reality exposure therapy gains be generalized to real-life? A meta-analysis of studies applying behavioral assessments. Behav Res Ther. 2015 Nov;74:18-24. doi: 10.1016/j.brat.2015.08.010. Epub 2015 Aug 31. PMID 26355646
- [Background] Schubert T, Friedmann F, Regenbrecht H. The experience of presence: Factor analytic insights. Presence: Teleoperators & Virtual Environments 10(3): 266-281, 2001.
- [Background] Steer RA, Brown GK, Beck AT, Sanderson WC. Mean Beck Depression Inventory-II scores by severity of major depressive episode. Psychol Rep. 2001 Jun;88(3 Pt 2):1075-6. doi: 10.2466/pr0.2001.88.3c.1075. PMID 11597055
- [Background] Vlemincx E, Van Diest I, De Peuter S, Bresseleers J, Bogaerts K, Fannes S, Li W, Van Den Bergh O. Why do you sigh? Sigh rate during induced stress and relief. Psychophysiology. 2009 Sep;46(5):1005-13. doi: 10.1111/j.1469-8986.2009.00842.x. Epub 2009 May 21. PMID 19497009
- [Background] Wilhelm FH, Gevirtz R, Roth WT. Respiratory dysregulation in anxiety, functional cardiac, and pain disorders. Assessment, phenomenology, and treatment. Behav Modif. 2001 Sep;25(4):513-45. doi: 10.1177/0145445501254003. PMID 11530714
- [Background] Wolitzky-Taylor KB, Horowitz JD, Powers MB, Telch MJ. Psychological approaches in the treatment of specific phobias: a meta-analysis. Clin Psychol Rev. 2008 Jul;28(6):1021-37. doi: 10.1016/j.cpr.2008.02.007. Epub 2008 Mar 7. PMID 18410984
- [Background] Wolpe J, Lazarus AA. Behavior therapy techniques: A guide to the treatment of neuroses.1966.